CLINICAL TRIAL: NCT06656195
Title: Comparison of Effect of Gluteus Maximus Strengthening and Hamstring Flexibility in Patients With Sacroiliac Joint
Brief Title: Comparison of Gluteus Maximus Strengthening and Hamstring Flexibility in Sacroiliac Joint Dysfinction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah IU Shanza kanwal
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Sacroiliac Dysfunction
Keywords: hamstring tightness; gluteus maximus strengthing; SIJ dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group A (Experimental): In week 1 SIJ Mobilization along with ,Single leg bridge ,alternating leg lifts ,clam Exercise,Prone hip extension with knee flexion. In week 2 SIJ Mobilization along with Side-squats,Star excursion exercise,Forward step-down.In week 3 SIJ Mobilization along with bilateral squat ,single leg squat ,split squat/lunge ,frontal step up ,lateral step up.In week 4 SIJ mobilization along with bilateral squat with a band and hip extension against resistance was done.Three times a week for 4 weeks In each session, a total of two sets of 12 repetitions each were carried out, with a 1 min rest time between sets.
  Interventions: Other: glueus maximus strengthening
- experimental group B (Active Comparator): SIJ mobilization and Soft tissue mobilization along with Static Hamstrings stretching (3 sets, 15 repetitions with a holding time of 15 seconds ,3 times a week for 4 week) and Dynamic hamstrings stretching(3 set, 15 repetitions with a holding time of 1 second, 3 times a week for 4 weeks.
  Interventions: Other: hamstring stretching group

INTERVENTIONS:
Other: glueus maximus strengthening — In week 1 SIJ Mobilization along with ,Single leg bridge ,alternating leg lifts ,clam Exercise,Prone hip extension with knee flexion. In week 2 SIJ Mobilization along with Side-squats,Star excursion exercise,Forward step-down.In week 3 SIJ Mobilization along with bilateral squat ,single leg squat ,split squat/lunge ,frontal step up ,lateral step up.In week 4 SIJ mobilization along with bilateral squat with a band and hip extension against resistance was done.Three times a week for 4 weeks In each session, a total of two sets of 12 repetitions each were carried out, with a 1 min rest time between sets.
  Arms: experimental group A
Other: hamstring stretching group — SIJ mobilization and Soft tissue mobilization along with Static Hamstrings stretching (3 sets, 15 repetitions with a holding time of 15 seconds ,3 times a week for 4 week) and Dynamic hamstrings stretching(3 set, 15 repetitions with a holding time of 1 second, 3 times a week for 4 weeks.
  Arms: experimental group B

SUMMARY:
The aim of this research is to compare effect of strengthening of gluteus maximus and hamstring flexibility on hamstring tightness in sacroiliac joint dysfunction.

DETAILED DESCRIPTION:
The sacroiliac joints (SIJ) are the largest diarthrodial auricular shape axial joints in the human body that connect the iliac bones to the sacrum. SIJ dysfunction is mostly caused by abnormal motion and misalignment of the joint. Worldwide, the prevalence of sacroiliac joint dysfunction (SIJD) lies within a range of 13% to 30%.In approximately 10% to 25% of patients; SIJD is a cause of mechanical low back and leg pain. Hamstrings muscle tightness is one of the major problems associated with SIJ dysfunction. Over- activation of the hip flexors and inhibition of the gluteus maximus are common in the hamstring tendinopathy patient population. With decreased gluteal activation, the hamstrings are dominant for hip extension and can lead to a repetitive stress on the fibers which would lead to its tendinopathy. GM contraction produces compression of the SI joint, and also contributes to the force transmission mechanism from the lower extremity to the pelvis through the SI joint during functional activities such as ambulation. Inappropriate timing of GM activation during gait is thought to be one of the causes of SIJ dysfunction, because it decreases shock absorption mechanism at the sacroiliac joint. Earlier onset of hamstrings activation has been noted in patients with SIJ dysfunction as compensation for delayed firing of the GM. Weakness of the GM also leads to slouched posture, makes walking extremely difficult, and necessitates substitution by hamstrings. Therefore, neuromuscular specific GM strengthening exercises reduce the forces going directly through the hamstring muscle and tendon and therefore protects it. Jennifer Saunders et al provides a linkage between mechanical dysfunction of the sacroiliac joint and alterations in muscle function around the pelvis which has the potential to lead to recurrent injuries of the hamstring muscles. Any injury that leads to abnormal movement of the sacroiliac joint can alter the information sent from mechanoreceptors receptors at the articular surface and this may explain the pattern of inhibition of the transversus abdominis, multifidus and ipsilateral gluteus maximus which is commonly reported with SIJ dysfunction. There is some evidence that hamstring spasm may accompany the dysfunction in a reflex attempt to stiffen the joint (force closure).

Conditions

Conditions: SIJ dysfunction

Keywords: hamstring tightness, strengthening of gluteus maximus, SIJ dysfunction Study Design Study Type: Interventional

Primary Purpose: Treatment

Study Phase: N/A

Interventional Study Model: N/A

Allocation: Randomize Enrollment: 44 [Actual]

Intervention After obtaining informed consent from participants, demographics will be recorded. Screening will be performed to assess health status. Participants will be educated about the procedure and significance of the test. Patients fulfilling the inclusion criteria will be randomized into 2 groups i.e. Group A, Group B and with the help of sealed envelope method. Patients in Group A will receive strength of Gluteus maximus. Group B will receive hamstring flexibility exercises.

Group A Group B Week 1 & 2

SIJ Mobilization

Week 1

* Single leg bridge
* alternating leg lifts
* clam Exercise
* Prone hip extension with knee flexion Week 2
* Side-squats
* Star excursion exercise
* Forward step-down
* TENS
* SIJ mobilization
* Soft tissue mobilization [17]
* Static Hamstrings stretching (3 sets, 15 repetitions with a holding time of 15 seconds ,3 times a week for 4 week)
* Dynamic hamstrings stretching (3 set, 15 repetitions with a holding time of 1 second, 3 times a week for 4 weeks [18].

Week 3 and 4 SIJ Mobilization

Week 3

* bilateral squat
* single leg squat
* split squat/lunge
* frontal step up
* lateral step up

Week 4:

* bilateral squat with a band
* hip extension against resistance.

(Three times a week for 4 weeks. In each session, a total of two sets of 12 repetitions each were carried out, with a 1 min rest time between sets) [16].

Outcome Measures

* . Active knee extension test The patient is positioned supine with the hip flexed 90 degrees (either actively or passively). The knee is then actively extended from a starting position of 90-degree flexion toward full extension. The test is positive for hamstring tightness if the angle of knee extension is greater than 20 degrees.
* Dynamometer It is a small device that the examiner holds against the patient's limb as the patient exerts a maximal force. Dynamometers measure the amount of force and shows on its screen.
* NPRS The NPRS is frequently employed to measure pain intensity, in which patients are asked to select a number (from 0 to 10) to represent their pain severity.
* Cluster of Laslett for Sacroiliac joint assessment:

The Cluster of Laslett is a tool used in SI joint assessment. Laslett proposes an algorithm comprising 4 provocative tests to identify the SI joint as the source of pain as the other two tests didn't have additional diagnostic value.

• Denver SI Joint Questionnaire Denver SI Joint Questionnaire is a brief, 10-question survey that assesses the impact of pain on daily life activities such as sitting, walking, getting up from chair, walking up and down the stairs, getting in and out of car, bending at the waist, kneeling, or squatting, lifting, sleeping, work, recreation, social life, sex life, or family/home activities, Joint Stability. For each question, there is a possible 5 points. Total score is calculated as (total scored/50) X 100%. Scores range from 0-100% with higher scores representing more disability.

Eligibility

Inclusion Criteria

* Both genders
* Patient with pain over the posterior aspect of SI joint
* Age between 25-45 years.
* Positive Active knee extension test (angle of knee extension greater than 20 degrees)
* Two of four test of Laslett cluster of Sacro-iliac dysfunction is positive.

Exclusion Criteria

* Herniated disc.
* Skin infection.
* Any contraindications for affected lower limb exercises (e.g., venous thrombosis, lymphedema).
* Patients with any post operative history of Hip joint fracture, subluxation, dislocation, diabetes, arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Patient with pain over the posterior aspect of SI joint
* Age between 25-45 years.
* Positive Active knee extension test (angle of knee extension greater than 20 degrees)
* Two of four test of Laslett cluster of Sacro-iliac dysfunction is positive.

Exclusion Criteria:

* Herniated disc.
* Skin infection.
* Any contraindications for affected lower limb exercises (e.g., venous thrombosis, lymphedema).
* Patients with any post operative history of Hip joint fracture, subluxation, dislocation, diabetes, arthritis.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Active knee extension test | baseline to 4th week
  It is use to measure hamstring flexibility.The patient is positioned supine with the hip flexed 90 degrees (either actively or passively). The knee is then actively extended from a starting position of 90-degree flexion toward full extension. The test is positive for hamstring tightness if the angle of knee extension is greater than 20 degrees.
Dynamometer | baseline to 4th week
  It. is used to measure strength .It is a small device that the examiner holds against the patient's limb as the patient exerts a maximal force. Dynamometers measure the amount of force and shows on its screen.

SECONDARY OUTCOMES:
NPRS | baseline to 4th week
  The NPRS is frequently employed to measure pain intensity, in which patients are asked to select a number (from 0 to 10) to represent their pain severity.
Denver SI Joint Questionnaire | baseline to 4th week
  Denver SI Joint Questionnaire is a brief, 10-question survey that assesses the impact of pain on daily life activities such as sitting, walking, getting up from chair, walking up and down the stairs, getting in and out of car, bending at the waist, kneeling, or squatting, lifting, sleeping, work, recreation, social life, sex life, or family/home activities, Joint Stability. For each question, there is a possible 5 points. Total score is calculated as (total scored/50) X 100%. Scores range from 0-100% with higher scores representing more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- DSK Rehab and physio, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No